CLINICAL TRIAL: NCT06457867
Title: Radiographic and Histomorphometric Assessment of Microfragmented Adipose Tissue Loaded on Bovine Graft on Ridge Preservation Versus Bovine Graft Only for Subsequent Implant Placement in the Maxillary Posterior Region, a Randomized Clinical Trial.
Brief Title: Assessment of Microfragmented Adipose Tissue Loaded on Bovine Graft Versus Bovine Graft Only on Ridge Preservation.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bashaer Maruf Jamaan Bayashot, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: microfragmented adipose tissue
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Tooth Mobility
Keywords: unrestorable caries lesions or affected periodontium.
MeSH Terms: conditions — Tooth Mobility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- microfragmented adipose tissue (Experimental): microfragmented adipose tissue loaded on bovine graft on ridge preservation
  Interventions: Procedure: microfragmented adipose tissue loaded on bovine graft
- bovine graft (Active Comparator): bovine graft only on ridge preservation
  Interventions: Procedure: microfragmented adipose tissue loaded on bovine graft

INTERVENTIONS:
Procedure: microfragmented adipose tissue loaded on bovine graft — microfragmented adipose tissue loaded on bovine graft on ridge preservation

SUMMARY:
Evaluation of maxillary alveolar ridge changes (bone quantity and quality as revealed by Radiographic and Histomorphometry) utilizing microfragmented adipose tissue loaded on bovine graft versus bovine graft only for maxillary posterior ridge preservation.

DETAILED DESCRIPTION:
All patients involved in this study will be divided into two groups; each group will receive a different graft of bone augmentation: Adipose tissue loaded on bovine graft will be utilized for the study group and bovine raft only for the control group.

After 6 months, patients will be evaluated histomorphometrically via core biopsy at the time of implant placement and radiographically via assessment of ridge height on CBCT.

Radiographic assessment that will be achieved by CBCT scan will be used to calculate the changes of bone height from base line (1week) to 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring implant treatment after tooth extraction due to either unrestorable caries lesions or affected periodontium.

  * Age group: above 21 years
  * Remaining natural teeth have good periodontal tissue support and occlusion showed sufficient inter arch space for future prosthesis.

Exclusion Criteria:

* General contraindications to implant surgery.

  * Subjected to irradiation in the head and neck area less than 1 year before implantation.
  * Poor oral hygiene and motivation.
  * Severe bruxism or clenching.
  * Systemic, immunologic, or debilitating diseases that could affect normal bone healing & local pathosis.
  * Treated or under treatment of intravenous amino bisphosphonates.
  * Active infection or severe inflammation in the area intended for implant placement.
  * Patients participating in other studies if the present protocol could not be properly followed.
  * Heavy smokers

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Quantity of bone (vertical bone height) | Quantity of bone (vertical bone height) by CBCT after 6 months
  By CBCT

SECONDARY OUTCOMES:
Quality of bone | Histological analysis (Core biopsy) Percentage of newly formed bone after 6 months
  Histological analysis (Core biopsy) Percentage of newly formed bone

IPD SHARING:
Plan to Share IPD: Yes
All patients involved in this study will be divided into two groups; each group will receive a different graft of bone augmentation: Adipose tissue loaded on bovine graft will be utilized for the study group and bovine raft only for the control group.
  For both groups: All Patients of both groups will be evaluated radiographically immediately and after 6 months post-operative by cone beam CT scan to record Alveolar ridge height.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After 6 months, patients will be evaluated histomorphometrically via core biopsy at the time of implant placement and radiographically via assessment of ridge height on CBCT.
  Radiographic assessment that will be achieved by CBCT scan will be used to calculate the changes of bone height from base line (1week) to 6 months postoperatively.